CLINICAL TRIAL: NCT06444217
Title: Gene Therapy Development and Validation for Huntington's Disease Fibro TG-HD
Acronym: FibroTG-HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-A00877-40
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: Huntington Disease
Keywords: Huntington; gene therapy; trans-splicing; fibroblasts
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Huntington's patient (Experimental): skin biopsy
  Interventions: Procedure: skin biopsy

INTERVENTIONS:
Procedure: skin biopsy — skin biopsy

SUMMARY:
Huntington's disease is a rare and fatal monogenic neurodegenerative disorder whose molecular origin is an expansion of CAG triplets within the first exon of the Huntingtin gene. Although a growing number of emerging therapies are in clinical trials, there are no proven neuroprotective or curative treatments approved by the health authorities, as they have not yet demonstrated any real therapeutic benefit or absence of toxicity. Trans-splicing gene therapy is defined as the correction of a mutated endogenous pre-messenger RNA by a therapeutic exogenous pre-messenger RNA. Trans-splicing is a suitable alternative approach, since it is capable of allelic selectivity and replacement of mutated sequences by the wild-type one, criteria that no therapy tested to date meets. This project involves the therapeutic validation of trans-splicing of Huntingtin gene transcripts, and will evaluate its therapeutic effects in vitro, into primary fibroblast cell lines derived from skin biopsies of Huntington's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 70 years.
* Signed written, free and informed consent to participate in the study.
* Patients with a CAG≥36 allele (with reduced or full penetrance). penetrance)
* People affiliated to or benefiting from a social security scheme.

Exclusion Criteria:

* Individuals who have participated in a gene therapy trial using AAV, ASO, mi/si/shRNA administration, likely to disrupt expression, splicing of pre-mRNAs, mRNA splicing, mRNA expression/regulation/translation, energy or protein metabolism directly or indirectly linked to the Huntingtin gene (HTT), its transcripts and proteins.
* Clinical or paraclinical elements that may suggest a differential diagnosis.
* People unable to express their consent.
* Pregnant, breast-feeding or parturient women
* People deprived of liberty by administrative or judicial decision
* People under legal protection (curatorship, guardianship).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2028-07-23 (Estimated)

PRIMARY OUTCOMES:
In vitro validation of a RNA trans-splicing gene therapy for the correction of supernumerary CAG repeats into fibroblasts derived from skin biopsies of patients with Huntington's disease. | At the inclusion
  Correction of mutated endogenous transcripts.

SECONDARY OUTCOMES:
Quantify the expression of Huntingtin protein (HTT) and its (in)usual protein partners. | At the inclusion
  At the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: VERNY Christophe, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- ABRIAL, Angers, Maine et Loire, France